CLINICAL TRIAL: NCT02094768
Title: Effects of Replacing Sugar Sweetened Beverages With Milk on Metabolic Factors in Overweight and Obese Adolescents
Brief Title: Soda and Milk Study
Acronym: SAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: MM7267
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Dyslipidemia
MeSH Terms: conditions — Obesity; Dyslipidemias | interventions — Diet, Fat-Restricted; Milk; Sugar-Sweetened Beverages

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reduced Fat Milk (Experimental): 20 oz. reduced fat (2%) milk per day
  Interventions: Dietary Supplement: Reduced Fat Milk
- Sugar Sweetened Soda (Experimental): 24oz. soda per day
  Interventions: Dietary Supplement: Sugar Sweetened Soda

INTERVENTIONS:
Dietary Supplement: Reduced Fat Milk — Subjects will be provided with and instructed to consume the equivalent of 20oz. reduced fat milk per day for 3 weeks
  Other Names: 2% milk
  Arms: Reduced Fat Milk
Dietary Supplement: Sugar Sweetened Soda — Subjects will be provided with and instructed to consume 2 cans (24oz) of sugar sweetened soda per day for 3 weeks
  Other Names: High fructose corn syrup sweetened soda
  Arms: Sugar Sweetened Soda

SUMMARY:
Much attention has been directed at the unhealthy effects of sugar-sweetened beverages (SSBs), as an increase in their consumption has paralleled the rise obesity rates. In adults, SSBs have been shown to promote ectopic fat storage and raise plasma triglycerides compared to equivalent amounts of semi-skim (1.5%) milk, water, or diet beverages. Replacement of soda with milk had the added benefit of also reducing systolic blood pressure. While several studies have investigated the effects of SSBs on weight gain in children, no published studies have investigated their effects on lipid and lipoprotein risk factors under isocaloric conditions in metabolically at-risk adolescents, who are among the greatest consumers of SSBs. The main objective of this study is to test whether isocaloric replacement of soda with reduced fat milk will significantly improve atherogenic dyslipidemia, blood pressure, insulin sensitivity, and liver function in overweight and obese adolescents who are habitual soda consumers. The investigators will test this in a 8 week randomized two period crossover trial in 30 overweight and obese adolescent males who are self-reported habitual consumers of SSBs. Participants will consume energy equivalent amounts of SSB (24oz soda containing high fructose corn syrup per day), and reduced fat milk (2% milk fat) for 3 weeks each, in random order, separated by a 2-week washout. Anthropometrics, blood pressure, and blood samples will be collected at screen and at the end of each intervention period. Plasma measurements will include LDL peak particle diameter; lipoprotein subclass concentrations; triglycerides; total, LDL, and HDL-cholesterol; apolipoproteins; glucose, insulin, and insulin resistance; high sensitivity C-reactive protein; uric acid; and liver enzymes.

ELIGIBILITY:
Inclusion Criteria:

* Males, age 13-18
* Tanner stage ≥ 2
* Self reported sugar sweetened beverage intake 24oz to 60oz per day
* Self reported milk intake ≤16 oz. per day
* BMI 85-99 percentile for age
* Tolerant to milk

Exclusion Criteria:

* History or diagnosis of hypertension or taking blood pressure lowering medication
* History or diagnosis of diabetes, HbA1c ≥ 6.5% or fasting glucose ≥ 126 mg/dl
* Fasting triglyceride > 300 mg/dl
* On lipid lowering or diabetes medication

Ages: 13 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
LDL peak particle diameter | 3 weeks

SECONDARY OUTCOMES:
Plasma triglycerides | 3 weeks
LDL-cholesterol | 3 weeks
HDL-cholesterol | 3 weeks
Blood pressure | 3 weeks
  Systolic and diastolic
LDL subclass concentrations | 3 weeks
Apolipoprotein B | 3 weeks
Apolipoprotein AI | 3 weeks
Apolipoprotein CIII | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Krauss, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Cholesterol Research Center, Berkeley, California, United States